CLINICAL TRIAL: NCT06066840
Title: Vedolizumab, Anti-CD25 Antibody Combined With Rapid Reduction of Glucocorticoids as Treatment of Grade 3-4 Steroid-resistant Acute Graft-versus-host Disease With Lower Gastrointestinal Involvement
Brief Title: Vedolizumab, Anti-CD25 Antibody, Rapid Reduction of Glucocorticoids for SR-aGVHD With Gastrointestinal Involvement
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GVHD002
Record Dates: First submitted 2023-07-31; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-04

CONDITIONS: Safety and Efficacy
MeSH Terms: interventions — Basiliximab; PC61 monoclonal antibody; vedolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- vedolizumab+basiliximab (Experimental): Patients with steroid-refractory aGVHD with gastrointestinal involvement receive combined therapy of vedolizumab and basiliximab.
  Interventions: Drug: Basiliximab; Drug: Vedolizumab

INTERVENTIONS:
Drug: Basiliximab — Basiliximab is a second-line treatment for steroid-resistant acute graft-versus-host disease.
  Other Names: anti-CD25 monoclonal antibody
Drug: Vedolizumab — Vedolizumab is a second-line treatment for steroid-resistant acute graft-versus-host disease.
  Other Names: anti-α4β7 monoclonal antibody

SUMMARY:
Acute graft-versus-host disease (aGVHD) is the most common life-threatening complication of allogeneic hematopoietic stem cell transplantation. The investigators try to observe the efficacy and safety of application of vedolizumab, anti-CD25 monoclonal antibody and rapid reduction of glucocorticoids in the treatment of grade 3-4 steroid-refractory aGVHD(SR-aGVHD) with lower gastrointestinal involvement.

DETAILED DESCRIPTION:
Sample size: According to Simon optimal two-stage design, P0=60%, P1=80%, α=0.05, β=0.2, a sample size of 45 was chosen.

Objects: Adults ages 18-65 diagnosed with grade 3-4 SR-aGVHD with lower gastrointestinal involvement.

Design

Participants with grade 3-4 SR-aGVHD with lower gastrointestinal involvement(progression after 3 days or lack of improvement after 5 days of 1-2 mg/kg/d systemic steroids) receive combined therapy of vedolizumab and anti-CD25 monoclonal antibody, with methylprednisolone terminated in 7-10 days.

Vedolizumab is given 300mg, day 1/15/43, and then once every 8 weeks until gastrointestinal GVHD reaches grade 1 (1 episodes for minimum).

Basiliximab is given 20mg twice a week for week 1, and then once a week until GVHD of the participants reaches grade 2(3 episodes for minimum). If basiliximab is not available, it can be replaced by recombinant humanized anti-CD25 monoclonal antibody injection, 50mg once with the same frequency.

Methylprednisolone is reduced to 1mg/kg/d at day 1 and is aborted in 7-10 days. If chronic GVHD or overlap syndrome is considered later during treatment, steroids (ie. methylprednisolone 0.5mg/kg/d) can be administered again.

Intravenous cyclosporine or tacrolimus is given and plasma concentration is monitored in a safe and effective range.

Best supportive treatment is given, including broad-spectrum anti-infection, nutrition support, and blood transfusion.

The investigators access the efficacy and safety of second-line therapy once a week from day 14 until complete remission is received. Then the investigators access the hematological disease status, aGVHD, cGVHD, infection state once a month.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of grade 3-4(according to MAGIC criteria) steroid-resistant acute graft-versus-host disease(progression after 3 days or lack of improvement after 5 days of systemic 1.5-2 mg/kg steroids) with gastrointestinal involvement.
* Age 18-65.
* ECOG score≤3.
* Must be able to understand and willing to participate in the study and sign the informed consent.

Exclusion Criteria:

* Refractory/secondary graft-versus-host disease.
* Severe complications such as myocardial infarction, chronic cardiac insufficiency,
* hepatic failure, renal insufficiency, etc.
* Clinically uncontrolled active infections.
* Other Malignant tumors with progression.
* Heart failure: EF<30%, NYHA≥grade III.
* Pregnant or lactating women.
* Expected survival <60 days.
* Undergoing other drug clinical trials.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
overall response rate at day 28 | day 28
  The primary endpoint is the overall response rate (ORR) at day 28 defined as proportion of patients demonstrating partial (PR) or complete response (CR) without requirement for additional systemic immunosuppressive therapy (IST) at day 28 after second-line treatment initiates.

SECONDARY OUTCOMES:
ORR at d14/d56 | day 14, day 56
  overall response rate at day 14/56
Duration of response | through study completion, an average of 1year
  Duration of response, assessed for responders only by calculating the time from first response to the date of first observation of aGvHD relapse/progression or the date of additional IST for GvHD.
OS | through study completion, an average of 1year
  Overall survival (OS) defined as time from the day treatment initiates to the date of death from any cause.
EFS | through study completion, an average of 1year
  Event-free survival (EFS) defined as the time from the day treatment initiates to the date of recurrence of underlying hematologic disease, graft failure or death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Xuefeng He, doctor, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No